CLINICAL TRIAL: NCT06940986
Title: The PROmoting Pain Self-Management (PROs) Trial: Holistic Pain Care in the Military Health System
Acronym: PROs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: 59th Medical Wing (U.S. Federal Agency); Desmond Doss Health Clinic, Schofield Barracks (Unknown); University of Utah (Other); Madigan Army Medical Center (U.S. Federal Agency); Bassett Army Community Hospital (Unknown); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Dan Rhon, Primary Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pending
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain; Musculoskeletal Pain; Musculoskeletal Pain Disorder
Keywords: Empowered Relief; Move to Health; Holistic Pain Care; stepped care; chronic musculoskeletal pain; self-management; pain management; military; holistic health
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Collagen Diseases; Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Empowered Relief (Active Comparator): Empowered Relief uses a single, 2-hour session to accomplish several key tasks including; pain education; experiential exercises; didactic content on pain responses, stress, and tension; techniques to affect the relaxation response; basic unhelpful thought restructuring; self-soothing actions; and completion of a per-sonalized self-management plan for empowered relief. Similar to CBT relaxation, ER participants receive a calming tool in the form of a binaural app. Unlike CBT, ER is mainly didactic, omits content such as activity planning and pacing, and is provided in a single session, eliminating ongoing therapeutic alliance and peer support.
  Interventions: Behavioral: Empowered Relief
- Move to Health (Active Comparator): Move to Health (M2H) is part of an initiative in the Military Health System to transform healthcare delivery with emphasis on the power of holistic care and self-management. M2H is operationalized using a health coaching model based on collaborative part-nership between patient and a trained coach to facilitate healthy behavior change. Health coaching is an evidence-based intervention for persons with chronic pain with improvements in physical activity, pain intensity and interference.
  Interventions: Behavioral: Move to Health
- Usual Care (Active Comparator): Usual care (UC) pain management will be provided at the discretion of the participant's primary care provider, consistent with a pragmatic clinical trial.
  Persons assigned to UC will be advised to follow the recommendations from their primary care provider and will be provided information about local resources at their respective Military Treatment Facility. The study team will not take additional steps to standardize or compel adherence to practice guidelines and will collect health care utilization outcomes through the the Millitary Health System Data Repository at the conclusion of the trial.
  Interventions: Other: Usual Care as determined by primary care provider

INTERVENTIONS:
Behavioral: Empowered Relief — ER is provided in a single, 2-hour session delivered remotely by trained instructors. ER has two main components: didactics and skills acquisition as outlined below. The ER class is administered virtually. The class includes the didactic and skill acquisition content. At the end of the class participants receive tangible items including the self-crafted, personalized catastrophizing cessation plan, a guided relaxation response audio file, and an electronic copy of the didactic class content.
  Arms: Empowered Relief
Behavioral: Move to Health — The M2H intervention is delivered virtually by trained health coaches using a 6-step process. The administration of M2H begins with an initial session with follow-up sessions scheduled every 1-2 weeks for up to 8 weeks or until the participant is ready to transition to self-management.
  Arms: Move to Health
Other: Usual Care as determined by primary care provider — Patients will receive care as determined by their primary care provider, with no input or control by the research team.
  Arms: Usual Care

SUMMARY:
The goal of this study is to improve pain care in the MHS by identifying effective, whole-person, non-pharmacologic interventions for persons with chronic musculoskeletal pain. The investigators will evaluate two promising, evidence-based holistic health interventions and compare them to usual care.

DETAILED DESCRIPTION:
Chronic pain is a ubiquitous problem and growing concern for the Military Health System (MHS). Chronic musculoskeletal (MSK) pain conditions are the most common chronic pain conditions in the MHS. Numerous recommendations have been made to improve care for chronic MSK pain in the MHS. First, the Office of the Army Surgeon General is promoting the transition of the MHS to a holistic health system that seeks to maintain, restore, and improve health through team-based care supporting self-management and recognizing the complex, biopsychosocial nature of chronic pain. Second, a stepped care approach to pain management is advocated to make less intense but effective, first-line care broadly available and to base subsequent care on response to first-line options. While the MHS has articulated its vision for holistic pain care delivered within a stepped care framework, there is a need for research addressing key questions of which interventions are most effective and how to operationalize the stepped care model. In addition, pragmatic, sustainable strategies to implement holistic pain care in the MHS are needed. Electronic health records (EHR) are increasingly used to implement evidence-based interventions, but have not been widely tested in the MHS. The MHS has deployed a new system-wide EHR with standards-based capabilities for decision-support, making EHR-based implementation a timely option with high potential for future scalability.

Design: Pragmatic, individually-randomized, type I hybrid effectiveness-implementation trial Methods: The investigators will use the EMR to help facilitate recruitment. The investigators plan to recruit a total of 608 persons with chronic MSK pain receiving care in the MHS. Participants providing consent will be randomized in 1 : 2.3 : 2.3 ratio to Usual Care (UC), Empowered Relief (ER), or Move to Health (M2H) for phase I treatment. All participants will be re-evaluated after 14 weeks. Participants initially assigned to the ER, determined to be non-responders to treatment, will receive M2H as a Phase II intervention to evaluate a stepped care process. All participants will also complete assessments at 26 and 52 weeks after randomization. The primary outcome will be a self-reported measure of pain impact. Secondary outcomes will include additional effectiveness measures. The research team will also evaluate implementation outcomes grounded in a Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework.

Summary: The goal of the promoting pain self-management (PROs) study is to improve pain care in the MHS by identifying effective, whole-person, non-pharmacologic interventions for persons with chronic MSK pain. The investigators plan to evaluate two promising, evidence-based interventions, ER and M2H, and also compare these to UC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* TRICARE Beneficiary
* Meets the case definition of chronic MSK pain requiring 2 or more medical encounters within the past year and at least 90 days apart for the same MSK condition indicated by medical encounter data or MSK pain ICD-10 codes in the electronic medical record

Exclusion Criteria:

* Actively receiving cancer treatment
* Currently known to be pregnant
* Receiving advanced chronic pain management, including multi-disciplinary or behavioral pain management or mental health or substance use programs (beyond the initial step of the VA/DoD stepped care model for pain management)
* Suicidal Ideation determined by a higher than lower risk score on the P4 Screener
* Currently undergoing post-surgical rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
3-PEG Scale | From enrollment to the end of treatment at 14 weeks
  The three items include 1 pain intensity item (Pain intensity during the past week) and 2 pain interference items (Pain interference with Enjoyment of life, and pain interference with General activity). The total score is the average of the three items (range, 0-10; higher scores indicate worse pain impact)

SECONDARY OUTCOMES:
PROMIS Physical Function | From enrollment to end of surveillance period at 52 weeks (including 14 and 26 week assessments)
  The PROMIS short form 6b for physical function uses fixed items from the PROMIS physical function item bank to provide a T-score with population mean = 50 (sd=10).96
PROMIS Sleep Disturbance | From enrollment to end of surveillance period at 52 weeks (including 14 and 26 week assessments)
  The PROMIS short form 6a for sleep disturbance uses fixed items from the PROMIS sleep disturbance item bank to provide a T-score with population mean = 50 (sd=10).
3-PEG Scale | From enrollment to the end of the surveillance period (26 and 52 weeks)
  The three items include 1 pain intensity item (Pain intensity during the past week) and 2 pain interference items (Pain interference with Enjoyment of life, and pain interference with General activity). The total score is the average of the three items (range, 0-10; higher scores indicate worse pain impact)
PROMIS Depression | From enrollment to end of surveillance period at 52 weeks (including 14 and 26 week assessments)
  The PROMIS short form 6a for depression uses fixed items from the PROMIS depression item bank to provide a T-score with population mean = 50 (sd=10).
PROMIS Fatigue | From enrollment to end of surveillance period at 52 weeks (including 14 and 26 week assessments)
  The PROMIS short form 6a for fatigue uses fixed items from the PROMIS fatigue item bank to provide a T-score with population mean = 50 (sd=10).
PROMIS Prescription Medication Misuse | From enrollment to end of surveillance period at 52 weeks (including 14 and 26 week assessments)
  The PROMIS short form 7a assesses the abuse of prescription pain medication over a 3-month period. The short form uses fixed items from the PROMIS item bank to provide a T-score with population mean = 50 (sd=10).
Sleep Duration | From enrollment to end of surveillance period at 52 weeks (including 14 and 26 week assessments)
  Sleep duration is assessed through a single item question that comes from the Pittsburgh Sleep Quality Index (PSQI): "During the past month, how many hours and minutes of actual sleep did you get at night? (This may be different than the number of hours and minutes you spent in bed)."
Pain Catastrophizing Scale (PCS) | From enrollment to end of surveillance period at 52 weeks (including 14 and 26 week assessments)
  The PCS is a 13-item scale assessing the extent to which people catastro-phize in response to pain. Each item is scored from 0-4 providing an overall score from 0-52.
Pain Self-Efficacy Scale (PSEQ) | From enrollment to end of surveillance period at 52 weeks (including 14 and 26 week assessments)
  The PSEQ is a 4-item scale assessing a person's confidence to achieve goals and perform activities even with pain. Each item is scored from 0-6 for an overall score ranging from 0-60.

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Fritz, PhD, Principal Investigator — University of Utah; Daniel I Rhon, PhD, Principal Investigator — Brooke Army Medical Center
Locations (5):
- United States (5):
  - Bassett Army Community Hospital, Fairbanks, Alaska
  - Desmond Doss Health Clinic, Schofield Barracks, Hawaii
  - Brooke Army Medical Center, San Antonio, Texas
  - Wilford Hall Ambulatory Surgical Center, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified demographic data (e.g., sex, age), and participant-reported outcomes data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be stored in a repository as required by the sponsor/funder (NCCIH).
Access Criteria: The public-use data files in this collection are available for access by the general public. Access does not require affiliation with an ICPSR member institution. Access to data is sometimes restricted and users are expected to adhere to norms for responsible use. Restricted data files are not available for direct download from the website. Users interested in obtaining these data must complete a Restricted Data Use Agreement, specify the reason for the request, and obtain IRB approval or notice of exemption for their research.
URL: https://www.icpsr.umich.edu/web/pages/

REFERENCES:
- [Background] Abiero B, Gliner M, Beamer S, Sackett A, Marshall-Aiyelawo K, Ellison J, McDavid T, de Geus J. Military Medical Readiness and Patient Experience with Access to Care. Med J (Ft Sam Houst Tex). 2022 Jan-Mar;(Per 22-01/02/03):3-10. PMID 34940962
- [Background] Adams RS, Thomas CP, Ritter GA, Lee S, Saadoun M, Williams TV, Larson MJ. Predictors of Postdeployment Prescription Opioid Receipt and Long-term Prescription Opioid Utilization Among Army Active Duty Soldiers. Mil Med. 2019 Jan 1;184(1-2):e101-e109. doi: 10.1093/milmed/usy162. PMID 30007291
- [Background] Institute of Medicine (US) Committee on Advancing Pain Research, Care, and Education. Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK91497/ PMID 22553896
- [Background] Department of Veterans Affairs. Veterans' Health Administration. Pain Management, VHA Directive 2009-053. October 28, 2009. Published 2009. Accessed August 25, 2023.
- [Background] Toblin RL, Quartana PJ, Riviere LA, Walper KC, Hoge CW. Chronic pain and opioid use in US soldiers after combat deployment. JAMA Intern Med. 2014 Aug;174(8):1400-1. doi: 10.1001/jamainternmed.2014.2726. No abstract available. PMID 24978399